CLINICAL TRIAL: NCT06434207
Title: Extracellular Vesicle Micro RNA Profiling in Congenital Heart Disease: Fetal-Maternal Regulation in Neonatal Thrombosis
Acronym: EVmiRNA
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Koichi Yuki, Principal Investigator, MD, Boston Children's Hospital
Other Study IDs: IRB-P00048093
Record Dates: First submitted 2024-05-12; First posted 2024-05-30 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-09

CONDITIONS: Congenital Heart Disease; Single-ventricle; Thrombosis
MeSH Terms: conditions — Heart Defects, Congenital; Univentricular Heart; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood from neonate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates with Congenital Heart Disease: Neonates born with severe Congenital Heart Disease undergoing corrective heart surgery within the first week of life under cardiopulmonary bypass at Boston Children's Hospital will be eligible for participation. As part of standard clinical care, neonates having cardiac surgery at Boston Children's Hospital have clinical labs drawn during and after surgery. All blood collected from neonates as part of this study will be discarded blood from those routine clinical samples. One sample will be taken before surgery and one sample will be taken after surgery.
  Interventions: Other: Collecting discarded blood samples

INTERVENTIONS:
Other: Collecting discarded blood samples — Discarded blood samples will be collected from routine clinical labs collected before and after surgery.

SUMMARY:
Newborns with congenital heart disease (CHD) are at increased risk of developing postpartum and postoperative blood clots after cardiac surgery. The molecular mechanisms that are responsible for the clotting profile predisposing children to blood clots in the early stages of life are currently not well described.

The goal of this proposal is to prospectively collect plasma samples from ten (10) neonates with antenatal diagnosis of severe congenital heart disease (CHD) to better understand mechanisms responsible for abnormal clotting in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* All neonates with a diagnosis of severe Congenital Heart Disease undergoing surgery at Boston Children's Hospital in the first week of life

Exclusion Criteria:

* None

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All neonates with a diagnosis of severe Congenital Heart Disease undergoing surgery at Boston Children's Hospital in the first week of life.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of microRNA in whole blood samples from neonates | 2 days
  isolation, purification and sequencing of patterns of miRNA and clustering analysis will be performed to determine predominant populations of miRNA related to inflammation, complement activation, and coagulation among other pathways

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States